CLINICAL TRIAL: NCT01581684
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 411034 (PIB) in Healthy Male Volunteers (Randomised, Single-blind, Placebocontrolled Within Dose Groups, Phase I Study)
Brief Title: Safety Tolerability and Pharmacokinetic of BI 411034
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1308.1; 2011-004840-23 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Healthy

ARMS (9):
- BI 411034 low dose - group 1 (Experimental): Solution for oral administration
  Interventions: Drug: BI 411034
- BI 411034 low dose - group 2 (Experimental): Solution for oral administration
  Interventions: Drug: BI 411034
- BI 411034 medium dose - group 3 (Experimental): Solution for oral administration
  Interventions: Drug: BI 411034
- BI 411034 medium dose - group 4 (Experimental): Solution for oral administration
  Interventions: Drug: BI 411034
- BI 411034 medium dose - group 5 (Experimental): Solution for oral administration
  Interventions: Drug: BI 411034
- BI 411034 high dose - group 6 (Experimental): Solution for oral administration
  Interventions: Drug: BI 411034
- BI 411034 high dose - group 7 (Experimental): Solution for oral administration
  Interventions: Drug: BI 411034
- BI 411034 high dose - group 8 (Experimental): Solution for oral administration
  Interventions: Drug: BI 411034
- Placebo (Placebo Comparator): Solution for oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 411034 — Low dose solution for oral administration
  Arms: BI 411034 low dose - group 2
Drug: Placebo — Solution for oral administration
  Arms: Placebo
Drug: BI 411034 — Medium dose solution for oral administration
  Arms: BI 411034 medium dose - group 3
Drug: BI 411034 — Low dose solution for oral administration
  Arms: BI 411034 low dose - group 1
Drug: BI 411034 — High dose solution for oral administration
  Arms: BI 411034 high dose - group 6
Drug: BI 411034 — High dose solution for oral administration
  Arms: BI 411034 high dose - group 7
Drug: BI 411034 — Medium dose solution for oral administration
  Arms: BI 411034 medium dose - group 5
Drug: BI 411034 — High dose solution for oral administration
  Arms: BI 411034 high dose - group 8
Drug: BI 411034 — Medium dose solution for oral administration
  Arms: BI 411034 medium dose - group 4

SUMMARY:
The primary objective of the current study is to investigate the safety, tolerability and pharmacokinetics of BI 411034 in healthy male volunteers following oral administration of single rising doses.

The secondary objective is to explore dose proportionality of BI 411034 in CYP2C19 (Cytochrome P450) genotyped extensive metabolisers (EM).

Another objective is to compare the safety and pharmacokinetic profiles between two different groups of CYP2C19 genotyped subjects, extensive metabolisers (EM) and poor metabolisers (PM)

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2012-08-01 (Actual); Study Completion 2012-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1308.1.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo EM: A powder for oral solution in the same volume as the respective active medication group and participants who are extensive metabolisers (EM)
- 2mg EM: Single oral dose of 2mg of BI 411034 for participants who are extensive metabolisers
- 8mg EM: Single oral dose of 8mg of BI 411034 for participants who are extensive metabolisers
- 20mg EM: Single oral dose of 20mg of BI 411034 for participants who are extensive metabolisers
- 40mg EM: Single oral dose of 40mg of BI 411034 for participants who are extensive metabolisers
- 80mg EM: Single oral dose of 80mg of BI 411034 for participants who are extensive metabolisers
- 150mg EM: Single oral dose of 150mg of BI 411034 for participants who are extensive metabolisers
- 250mg EM: Single oral dose of 250mg of BI 411034 for participants who are extensive metabolisers
- Placebo PM: A powder for oral solution in the same volume as the respective active medication group and participants who are poor metabolisers (PM)
- 20/60mg PM: Single oral dose of 20/60mg of BI 411034 for participants who are poor metabolisers
Period: Overall Study
Arm/Group | Placebo EM | 2mg EM | 8mg EM | 20mg EM | 40mg EM | 80mg EM | 150mg EM | 250mg EM | Placebo PM | 20/60mg PM
Started | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1 | 5
Completed | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other reason not defined | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo EM | 2mg EM | 8mg EM | 20mg EM | 40mg EM | 80mg EM | 150mg EM | 250mg EM | Placebo PM | 20/60mg PM | Total
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1 | 5 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (6.3) | 35.5 (9.9) | 39.8 (4.3) | 38.8 (8.7) | 38.3 (8.2) | 39.5 (3.1) | 32.7 (5.4) | 43.8 (6.7) | 31.0 (NA) — Measure of dispersion not possible to calculated for one participant | 42.4 (8.6) | 38.6 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1 | 5 | 62

OUTCOME MEASURES:

1. Secondary Outcome: Maximum Measured Concentration (Cmax )
Description: Maximum measured concentration of the analyte (BI 411034) in plasma
Time Frame: 2 hours (h) before drug administration and 10 minutes (min), 20min, 30min, 45min, 1h 15min, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 48h, and 72h after drug administration
Population: PK analysis set which included all subjects who were administered trial medication and were documented to have taken the dose of investigational treatment and who provided at least one observation for at least one pharmacokinetic (PK) endpoint without important protocol violations relevant to the evaluation of PK
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- 20mg PM: Single oral dose of 20mg of BI 411034 for participants who are poor metabolisers
- 60mg PM: Single oral dose of 60mg of BI 411034 for participants who are poor metabolisers
Arm/Group | 2mg EM | 8mg EM | 20mg EM | 40mg EM | 80mg EM | 150mg EM | 250mg EM | 20mg PM | 60mg PM
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
nmol/L | 61.7 (34.0) | 236 (55.9) | 566 (22.0) | 629 (53.9) | 2630 (38.8) | 4610 (51.4) | 6600 (15.3) | 935 (17.1) | 2890 (36.5)

2. Secondary Outcome: Time to Maximum Measured Concentration (Tmax)
Description: Time from dosing to maximum measured concentration
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Median (Full Range); unit: h
Arm/Group | 2mg EM | 8mg EM | 20mg EM | 40mg EM | 80mg EM | 150mg EM | 250mg EM | 20mg PM | 60mg PM
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
h | 0.5 [0.5 to 0.52] | 0.63 [0.48 to 1.50] | 0.63 [0.50 to 1.00] | 1.00 [0.75 to 1.50] | 0.62 [0.33 to 0.75] | 0.62 [0.48 to 1.02] | 0.63 [0.50 to 0.77] | 0.75 [0.50 to 1.00] | 0.50 [0.33 to 3.00]

3. Secondary Outcome: Area Under the Curve From 0 Extrapolated to Infinity (AUC0-infinity)
Description: Area under the concentration-time curve of the analyte (BI 411034) in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 2mg EM | 8mg EM | 20mg EM | 40mg EM | 80mg EM | 150mg EM | 250mg EM | 20mg PM | 60mg PM
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
nmol*h/L | 134 (54.3) | 729 (96.4) | 1410 (18.1) | 1900 (66.2) | 6140 (53.6) | 13300 (70.6) | 19700 (47.7) | 6240 (14.8) | 18500 (13.1)

4. Secondary Outcome: Amount of Analyte Eliminated in Urine From 0h to 4h (Ae0-4)
Description: Amount of analyte (BI 411034) eliminated in urine from the time point 0h to time point 4h.
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol
Arm/Group | 2mg EM | 8mg EM | 20mg EM | 40mg EM | 80mg EM | 150mg EM | 250mg EM | 20mg PM | 60mg PM
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
nmol | 77.6 (50.3) | 290 (22.1) | 530 (38.2) | 860 (34.1) | 2070 (38.8) | 3390 (44.6) | 4520 (25.9) | 1220 (30.3) | 3080 (22.1)

5. Primary Outcome: Number of Participants With Drug Related AEs
Description: Number of participants with drug related adverse events (AEs)
Time Frame: From drug administration until end of trial examination, up to 13 days
Population: Treated set which included all subjects who were administered trial medication and were documented to have taken the dose of investigational treatment
Measure: Number; unit: participants
Arm/Group | Placebo EM | 2mg EM | 8mg EM | 20mg EM | 40mg EM | 80mg EM | 150mg EM | 250mg EM | Placebo PM | 20mg PM | 60mg PM
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1 | 5 | 5
participants | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 3 | 0 | 0 | 2

6. Primary Outcome: Clinically Relevant Abnormalities for Physical Examinations, Vital Signs, ECG, Laboratory Tests
Description: Clinically relevant abnormalities for physical examinations, vital signs (blood pressure, pulse rate, oral body temperature, orthostasis test), 12-lead electrocardiogram (ECG) and clinical laboratory tests. Clinically relevant abnormalities are reported by the investigator as adverse events (AEs).
Time Frame: From drug administration until end of trial examination, up to 13 days
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Placebo EM | 2mg EM | 8mg EM | 20mg EM | 40mg EM | 80mg EM | 150mg EM | 250mg EM | Placebo PM | 20mg PM | 60mg PM
Number analyzed (Participants) | 14 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 1 | 5 | 5
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From drug administration until end of trial examination, up to 13 days
Arm/Group | Placebo EM | 2mg EM | 8mg EM | 20mg EM | 40mg EM | 80mg EM | 150mg EM | 250mg EM | Placebo PM | 20mg PM | 60mg PM
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/1 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/14 | 0/6 | 1/6 | 1/6 | 1/6 | 2/6 | 2/6 | 3/6 | 1/1 | 0/5 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo EM (N=14) | 2mg EM (N=6) | 8mg EM (N=6) | 20mg EM (N=6) | 40mg EM (N=6) | 80mg EM (N=6) | 150mg EM (N=6) | 250mg EM (N=6) | Placebo PM (N=1) | 20mg PM (N=5) | 60mg PM (N=5)
Chromatopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeling drunk (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 1
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes